CLINICAL TRIAL: NCT04424446
Title: Evaluation of Saliva as Source of Detection for SARS-CoV-2
Brief Title: Saliva as Source of Detection for SARS-CoV-2
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 200128; 20-CC-0128
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
Keywords: Coronavirus; COVID-19; SARS-CoV-2 RT-PCR; Severe Acute Respiratory Syndrome Coronavirus 2
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- NIH staff: NIH staff undergoing standard NIH COVID-19 screening willing to donate additional research samples.

SUMMARY:
Background:

Nasopharyngeal (NP) swabbing is being used to test for SARS-CoV-2 infection. For this, a swab is inserted deep into the back of the nose to collect a sample. It can cause discomfort for most people. Researchers want to find an easier way to collect samples.

Objective:

To learn if testing for SARSCoV-2 with a saliva sample only, a nasal swab from just the front part of the nostril only, or a saliva sample plus a nasal swab gives results that are as accurate as the NP swab.

Eligibility:

NIH staff members age 18 and older who are taking part in NIH CC SARS-CoV-2 surveillance.

Design:

The Occupational Medical Service (OMS) collects NP swabs as part of standard NIH staff screening. Participants will give 1 or 2 saliva samples and 1 or 2 nasal swabs when their NP swab is collected by OMS. If their NP swab was already collected, their OMS record will be reviewed for the result.

If the NP swab result is positive, the participant will have another NP swab. At that time, they will also give 1 or 2 saliva samples and 1 or 2 nasal swabs. If the NP swab result is negative, they will give 1 or 2 saliva samples and 1 or 2 nasal swabs the next time they have an NP swab.

For the saliva sample, participants will spit into a tube.

For the nasal swab, the inside of the front part of the nostril will be swabbed.

Participation ends after the study samples are collected. Participants can choose to keep giving saliva and nasal swab samples each time they have an NP swab.

DETAILED DESCRIPTION:
Because of the inconvenience of nasopharyngeal (NP) testing for SARS-CoV-2 detection, we are interested in identifying different strategies for detecting infection. A technique that is less intrusive would put individuals undergoing testing at lower risk for complications, would likely increase compliance with subsequent tests, and would decrease risk to the providers who are conducting the test. For asymptomatic screening, some institutions are using midturbinate swabs instead of NP swabs, for increased compliance due to decreased discomfort. The NIH has switched to midturbinate collection in asymptomatic collections only. A test that would require only expectorating saliva and/or collection of a midturbinate swab would address the issues of NP collection discomfort. Saliva is the most preferred by patients or asymptomatic staff due to no collection in the nasal cavity at all. Although the CDC lists midturbinate swab as an acceptable specimen type, there are minimal data about the sensitivity of this collection for SARS-CoV-2, and decisions to use midturbinate swabs are based in part on experience with other respiratory viruses. Also, if saliva were found to be equivalent to NP for patient testing, there will be a benefit to future patients in providing this option for testing. Therefore, we propose to validate these sample types for SARS-CoV-2 detection. The RT-PCR results based on a saliva sample alone or a saliva sample coupled with a midturbinate swab, will be correlated with the results using surveillance or diagnostic swab samples to validate their use for SARS-CoV-2 detection.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Is one of the following:

   1. An NIH staff member participating in NIH CC SARS-CoV-2 surveillance, or
   2. A WHC patient who had or is having a diagnostic NP RT-PCR test for SARS-CoV-2.
2. Age greater than or equal to 18 years.
3. Able to provide informed consent.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Inability or unwillingness to have NP sampling or midturbinate sampling (applies to NIH site only).
2. Inability or unwillingness to provide saliva sample (applies to both NIH and WHC sites).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NIH staff undergoing standard NIH COVID-19 screening
Sampling Method: Non-Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Saliva SARS-CoV-2 RT-PCR test results | Screening
  Validate saliva or nasal swab as a source of detection for SARS-CoV-2.

SECONDARY OUTCOMES:
Saliva and midturbinate swab SARS-CoV-2 RT-PCR test results | Screening
  Validate saliva coupled with a nasal swab as a source of detection for SARS-CoV-2.

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Frank, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (2):
- United States (2):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-CC-0128.html